CLINICAL TRIAL: NCT03322969
Title: Receiving Modified Chemotherapy Followed With Radical Resection After Neoadjuvant Chemotherapy Versus Receiving the Original Chemotherapy in Locally Advanced Gastric Cancer: a Randomized Controlled Study
Brief Title: Receiving Modified Chemotherapy Followed With Radical Resection After Neoadjuvant Chemotherapy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NAC-GC
Record Dates: First submitted 2017-10-24; First posted 2017-10-26 (Actual); Last update posted 2021-02-26 (Actual); Status verified 2021-02

CONDITIONS: Locally Advanced Gastric Cancer

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- receiving modified chemotherapy (Experimental): Paclitaxel/DDP
  Interventions: Drug: Paclitaxel/DDP
- receiving the original chemotherapy (Active Comparator): XELOX/SOX
  Interventions: Drug: XELOX/SOX

INTERVENTIONS:
Drug: Paclitaxel/DDP — receiving the modified chemotherapy
  Other Names: Group A
  Arms: receiving modified chemotherapy
Drug: XELOX/SOX — receiving the original chemotherapy
  Other Names: Group B
  Arms: receiving the original chemotherapy

SUMMARY:
For patients undergoing postoperative therapy for locally advanced gastric cancer after neoadjuvant chemotherapy, we assessed the utility of graded histologic regression of <50% as the criterion of treatment change. Sixty patients will be enrolled to randomize into two groups：receiving modified chemotherapy and receiving the original chemotherapy.

DETAILED DESCRIPTION:
For patients undergoing postoperative therapy for locally advanced gastric cancer after neoadjuvant chemotherapy, we assessed the utility of graded histologic regression of <50% as the criterion of treatment change. Sixty patients will be enrolled to randomize into two groups：receiving modified chemotherapy and receiving the original chemotherapy. Overall survival and disease-free survival will be observed between two groups.

ELIGIBILITY:
Inclusion Criteria:

* TNM stage of T2-T4 or positive regional lymph nodes, according to the American Joint Committee on Cancer (AJCC) 7.0 staging system, verified by enhanced abdominal computed tomography (CT) and/or endoscopic ultrasound (EUS), positron emission tomography (PET)/CT scan), with no evidence of distant metastases;
* ECOG performance status score ≤2 without serious heart, lung, liver, kidney, or hematological dysfunctions;
* age ≥18 years old;
* no previous chemotherapy, radiotherapy, or surgical treatment for gastric cancer;
* gastrectomy was performed after preoperative chemotherapy if imaging studies did not confirm disease progression (according to the Response Evaluation Criteria in Solid Tumors (RECIST)) ;
* signed the informed consent form.

Exclusion Criteria:

* All do not reach the inclusion criteria

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-08-23 (Actual); Primary Completion 2022-08 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
disease free survival | 3 year
  DFS between two arms

CONTACTS AND LOCATIONS:
Overall Officials: Lin Zhao, Doctor, Study Director — Department of Medical Oncology, Peking Union Medical College Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Department of Medical Oncology, Peking Union Medical College Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No